CLINICAL TRIAL: NCT01955330
Title: Long Term Follow-up of Robotic Hybrid Surgical Revascularization With CT Angiography
Brief Title: Long Term Follow-up Hybrid Revascularization
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: London Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: Kiaii-LTFUP-Hybrid-2013; REB #15000 (Other: Lawson Health Research Institute)
Record Dates: First submitted 2013-09-27; First posted 2013-10-07 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Coronary Artery Disease
Keywords: CABG, Hybrid, Robotic surgery
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hybrid robotic cabg patients: Postoperative (5-7 years)Hybrid CABG robotically assisted surgical revascularization patients
  Interventions: Procedure: Robotic Hybrid coronary artery revascularization

INTERVENTIONS:
Procedure: Robotic Hybrid coronary artery revascularization — Lita to LAD performed by robot, Hybrid stent to other diseased coronary artery
  Other Names: Robotic Hybrid CABG

SUMMARY:
OBJECTIVES:

The objectives of the year study are two-fold:

1. To determine the 5-7 year patency rate (rate of open bypass grafts) of the LITA graft and stent of patients who have already had robotically-assisted Hybrid CABG surgery using CTA and MPS-MIBI.
2. To determine patient quality of life at 5-7 years after robotically-assisted Hybrid CABG surgery

DETAILED DESCRIPTION:
New techniques such as robotically-assisted Hybrid CABG surgery need proper evaluation to ensure potential benefits gained are not harmful to that which we know to be of significant benefit to the patients, that being the left internal thoracic artery (LITA) graft (one of the main coronary arteries supplying your heart with blood). We are therefore proposing a 5-7 year CT-Angiography (CTA) and Myocardial Perfusion Scintigraphy (MPS-MIBI) to assess the patency rate of the LITA graft and the stented graft in patients that have already undergone robotically assisted Hybrid CABG.

ELIGIBILITY:
Inclusion Criteria:

- Patients that have previously had Hybrid robotic coronary artery revascularization performed approximately 5-7 years ago at the London Health Sciences Centre, University Hospital by Dr. Kiaii.

Exclusion Criteria:

- Patients not described above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have previously had Hybrid robotic coronary artery revascularization performed approximately 5-7 years ago at the London Health Sciences Centre, University Hospital by Dr. Kiaii.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Graft patency | 5-7 years post Hybrid surgery
  To assess the graft patency of the LITA to LAD performed by the robot and the patency of the Stent.

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, University & Victoria Hospitals, London, Ontario, Canada